CLINICAL TRIAL: NCT06474988
Title: Characterization of Biophysical and Mechanical Parameters on the Skin of Subjects With a Diagnosis of Breast Cancer After Surgery and Undergoing Adjuvant Treatment.
Brief Title: Characterization of Biophysical and Mechanical Parameters on Skin of Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: L2-094
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Estrogen Receptor Positive Tumor
Keywords: Estrogen Receptor Positive Breast Cancer; Adjuvant Treatment; Skin Toxicity
MeSH Terms: conditions — Breast Neoplasms | interventions — Skin Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tamoxifen: Patients who are receiving treatment with tamoxifen in adjuvant setting
  Interventions: Other: Skin tests
- Aromatase Inhibitors: Patients who are receiving treatment with an aromatase inhibitor in adjuvant setting
  Interventions: Other: Skin tests
- Paclitaxel: Patients who are receiving treatment with Paclitaxel in adjuvant setting
  Interventions: Other: Skin tests

INTERVENTIONS:
Other: Skin tests — Acquisition of Skindex questionnaire 29 and execution of instrumental skin tests

SUMMARY:
Aim of this study is to characterize the chemical/physical and structural parameters of the skin in patients with breast cancer undergoing oncological adjuvant treatment in order to understand how to prevent and manage adverse skin events during hormone therapy, also through the formulation of new functional dermocosmetics.

DETAILED DESCRIPTION:
Breast cancer is the most frequent neoplasm in women in industrialized countries. After surgery, an adjuvant systemic treatment is generally proposed (hormone therapy, chemotherapy, molecular targeted therapy).

Side effects of endocrine treatments, including skin toxicities, are frequent and often underestimated, leading to poor treatment adherence that can compromise therapeutic outcomes. Among adjuvant chemotherapy treatments, one of the most used drug is Paclitaxel: at skin level it can induce rash, dry skin and itching.

The combination of radiotherapy with these oncological treatments could aggravate cutaneous side effects.

Aim of this study is to characterize the chemical/physical and structural parameters of the skin in patints with breast cancer undergoing adjuvant treatment, performing specific skin tests with professional instruments and adequate personnel. The evaluation will be carried out in Estrogen Receptor (ER) positive breast cancer patients undergoing adjuvant therapy with Tamoxifen or Aromatase Inhibitor or Paclitaxel +/- adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age between 40 and 70 years
* subjects who are receiving treatment with tamoxifen, aromatase inhibitor or paclitaxel in adjuvant therapy +/- adjuvant radiotherapy
* subjects who are receiving hormonal therapy must have suspended any chemotherapy for at least 30 days

Exclusion Criteria:

* presence of known chronic skin pathologies before adjuvant treatment start (psoriasis, lupus, atopic dermatitis)
* inability to understand and will
* unavailability to carry out all the tests required by the protocol

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Estrogen receptor (ER) positive breast cancer patients undergoing adjuvant therapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Forearm hydration degree assessmnent | 1 day
  Forearm hydration degree evaluated using instrumental skin tests
Evaluation of Effects of Skin Disease on Quality of Life | 1 day
  Collection of Skindex29 questionnaire (minimum value: 1, maximum value: 5 - higher scores mean a greater agreement with the statement)

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Tosti, MD, Principal Investigator — European Istitute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy